CLINICAL TRIAL: NCT02376699
Title: A Phase 1, Open-label, Dose-escalation Study of SEA-CD40 in Adult Patients With Advanced Malignancies
Brief Title: Safety Study of SEA-CD40 in Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed due to portfolio prioritization
Sponsor: Seagen Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGNS40-001; PN 863 (Other: Merck Sharp & Dohme Corp)
Record Dates: First submitted 2015-02-17; First posted 2015-03-03 (Estimated); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell; Hodgkin Disease; Lymphoma; Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Melanoma; Neoplasm Metastasis; Neoplasms, Head and Neck; Neoplasms, Squamous Cell; Non-Small Cell Lung Cancer; Non-Small Cell Lung Cancer Metastatic; Non-small Cell Carcinoma; Squamous Cell Cancer; Squamous Cell Carcinoma; Squamous Cell Carcinoma of the Head and Neck; Squamous Cell Neoplasm; Lymphoma, Non-Hodgkin; Pancreatic Adenocarcinoma
Keywords: CD40 Antigen; Drug Therapy; Follicular Lymphoma; Hodgkin Disease; Immunotherapy; Indolent Lymphoma; Lymphoma; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Monoclonal Antibody; Neoplasms; Neoplasm Metastasis; Solid tumor; Seattle Genetics
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell; Hodgkin Disease; Lymphoma; Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Melanoma; Neoplasm Metastasis; Head and Neck Neoplasms; Neoplasms, Squamous Cell; Squamous Cell Carcinoma of Head and Neck; Lymphoma, Non-Hodgkin; Neoplasms | interventions — pembrolizumab; Injections, Subcutaneous; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- IV Monotherapy in Solid Tumors (Experimental): SEA-CD40 administered IV
  Interventions: Drug: Intravenous (IV) SEA-CD40
- IV Monotherapy in Lymphomas (Experimental): SEA-CD40 administered IV
  Interventions: Drug: Intravenous (IV) SEA-CD40
- Combination Therapy in Solid Tumors (Experimental): SEA-CD40 (administered IV) + pembrolizumab
  Interventions: Drug: Intravenous (IV) SEA-CD40; Drug: Pembrolizumab
- SC Monotherapy in Solid Tumors (Experimental): SEA-CD40 administered SC
  Interventions: Drug: Subcutaneous (SC) SEA-CD40
- SC Monotherapy in Lymphomas (Experimental): SEA-CD40 administered SC
  Interventions: Drug: Subcutaneous (SC) SEA-CD40
- Combination Therapy in Pancreatic Cancer (Experimental): SEA-CD40 (administered IV) + pembrolizumab + gemcitabine + nab-paclitaxel
  Interventions: Drug: Intravenous (IV) SEA-CD40; Drug: Pembrolizumab; Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Intravenous (IV) SEA-CD40 — Given intravenously; schedule is cohort-specific.
  Other Names: SEA-CD40
  Arms: Combination Therapy in Pancreatic Cancer; Combination Therapy in Solid Tumors; IV Monotherapy in Lymphomas; IV Monotherapy in Solid Tumors
Drug: Pembrolizumab — Given intravenously; schedule is cohort-specific.
  Other Names: Keytruda
  Arms: Combination Therapy in Pancreatic Cancer; Combination Therapy in Solid Tumors
Drug: Subcutaneous (SC) SEA-CD40 — Given subcutaneously on Day 1 every 3 weeks
  Other Names: SEA-CD40
  Arms: SC Monotherapy in Lymphomas; SC Monotherapy in Solid Tumors
Drug: Gemcitabine — 1000 mg/m^2 given intravenously on Day 1, 8, and 15 of each 28-day cycle
  Other Names: Gemzar
  Arms: Combination Therapy in Pancreatic Cancer
Drug: Nab-paclitaxel — 125 mg/m^2 given intravenously on Day 1, 8, and 15 of each 28-day cycle
  Other Names: Abraxane
  Arms: Combination Therapy in Pancreatic Cancer

SUMMARY:
This study is being done to find out if SEA-CD40 is safe and effective when given alone, in combination with pembrolizumab, and in combination with pembrolizumab, gemcitabine, and nab-paclitaxel. The study will test increasing doses of SEA-CD40 given at least every 3 weeks to small groups of patients. The goal is to find the highest dose of SEA-CD40 that can be given to patients that does not cause unacceptable side effects. Different dose regimens will be evaluated. Different methods of administration may be evaluated. The pharmacokinetics, pharmacodynamic effects, biomarkers of response, and antitumor activity of SEA-CD40 will also be evaluated.

DETAILED DESCRIPTION:
The study will be conducted in the following parts:

Part A: Intravenous (IV) monotherapy dose-regimen finding for solid tumors -- Dose-escalation, and possible dose-interval modification to lengthen the treatment cycle, to define the IV SEA-CD40 monotherapy maximum tolerated dose (MTD) and/or the optimal biological dose (OBD) regimens in patients with solid tumors. The ability to increase the dose intensity (to give additional doses within a treatment cycle) may be evaluated.

Part B: IV monotherapy solid tumor expansion cohorts -- Disease-specific solid tumor expansion cohorts may be enrolled where patients will be treated with doses at or below the IV SEA-CD40 monotherapy MTD and/or OBD determined in Part A.

Part C: IV monotherapy dose-regimen finding for lymphomas -- Dose-escalation, and possible dose-interval modification to lengthen the treatment cycle, to define the IV SEA-CD40 monotherapy MTD and/or the OBD regimens in patients with lymphomas. The ability to increase the dose intensity (to give additional doses within a treatment cycle) may be evaluated.

Part D: IV monotherapy lymphoma expansion cohorts -- Disease-specific lymphoma expansion cohorts may be enrolled where patients will be treated with doses at or below the IV SEA-CD40 monotherapy MTD and/or OBD determined in Part C.

Part E: Combination therapy dose-regimen finding for solid tumors -- IV SEA-CD40 dose-escalation to define the MTD and/or the OBD regimen to be administered in combination with standard approved dose of pembrolizumab in patients with solid tumors.

Part F: Combination therapy solid tumor expansion cohorts -- Disease-specific solid tumor expansion cohorts may be enrolled where patients will be treated with IV SEA-CD40 and pembrolizumab combination therapy; doses of SEA-CD40 will be at or below the MTD and/or OBD determined in Part E.

Part G: Subcutaneous (SC) injection (injected under the skin) monotherapy dose-regimen finding for solid tumors -- Dose-escalation, and possible dose-interval modification to lengthen the treatment cycle, to define the SC SEA-CD40 monotherapy maximum tolerated dose (MTD) and/or the optimal biological dose (OBD) regimens in patients with solid tumors.

Part H: SC monotherapy solid tumor expansion cohorts -- Disease-specific solid tumor expansion cohorts may be enrolled where patients will be treated with doses at or below the SC SEA-CD40 monotherapy MTD and/or OBD determined in Part G.

(Note: There is no Part I)

Part J: SC monotherapy dose-regimen finding for lymphomas -- Dose-escalation, and possible dose-interval modification to lengthen the treatment cycle, to define the SC SEA-CD40 monotherapy MTD and/or the OBD regimens in patients with lymphomas.

Part K: SC monotherapy lymphoma expansion cohorts -- Disease-specific lymphoma expansion cohorts may be enrolled where patients will be treated with doses at or below the SC SEA-CD40 monotherapy MTD and/or OBD determined in Part J.

Part L: Combination therapy in pancreatic cancer -- Patients will be treated with SEA-CD40 doses at or below MTD and/or OBD. An established dose of pembrolizumab and a standard regimen of gemcitabine and nab-paclitaxel will be used.

In Parts A, C, E, G, and J, a maximum feasible dose (MFD) will be defined if an MTD and/or OBD cannot be identified. Parts B, D, F, H, K. and L will explore the recommended dosing regimen once the MTD and/or OBD, or MFD (if the MTD and/or OBD cannot be identified) has been determined.

ELIGIBILITY:
Inclusion Criteria:

* (Monotherapy - Parts A, B, C, D, G, H, J, and K) -- Histologically confirmed advanced malignancy, either: (a) Metastatic or unresectable solid malignancy; or (b) Classical Hodgkin lymphoma (HL), or diffuse large B-cell lymphoma (DLBCL), or indolent lymphoma (including follicular lymphoma [FL])
* (Monotherapy - Parts A, B, C, D, G, H, J, and K) -- Relapsed, refractory, or progressive disease, specifically: (a) Solid tumors: Following at least 1 prior systemic therapy, and no further standard therapy is available for the patient's advanced solid tumor at the time of enrollment; or (b) Classical HL: Following at least 2 prior systemic therapies in patients who are not candidates for autologous stem cell transplant (SCT), or following failure of autologous SCT; or (c) DLBCL: Following at least 1 prior systemic therapy; patients must have also received intensive salvage therapy unless they refused or were deemed ineligible; or (d) Indolent lymphoma: Following at least 1 prior chemoimmunotherapy regimen that included an anti-CD20 monoclonal antibody and for which no other more appropriate treatment option exists
* (Combination Therapy - Part E and Part F) -- Histologically or cytologically confirmed advanced or metastatic solid malignancy for which pembrolizumab treatment is approved. In Part F, other advanced solid tumor indications may be eligible as identified by the Sponsor.
* (Pancreatic Cancer Cohort - Part L) - Histologically or cytologically confirmed metastatic exocrine ductal adenocarcinoma of the pancreas not amenable to curative therapy. Patients must not have received any prior systemic therapy for metastatic disease; patients who have received prior therapy for non-metastatic pancreatic adenocarcinoma are eligible if therapy was fully completed more than 4 months before start of study treatment.
* Representative baseline tumor tissue sample is available (Parts A-K)
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate baseline hematologic, renal, and hepatic function
* Recovery to Grade 1 of any clinically significant toxicity attributed to prior anticancer therapy prior to initiation of study drug administration

Exclusion Criteria:

* Parts A-K

  1. Prior chemotherapy, small molecule inhibitors, and/or other investigational anticancer agents (excluding investigational monoclonal antibodies) within 4 weeks
  2. Prior radiotherapy: therapeutic radiotherapy within 4 weeks, or palliative radiotherapy (to non-CNS disease) within 1 week
  3. Prior immune-checkpoint inhibitors within 4 weeks (or 8 weeks, if immuno-oncology doublet used as the prior line of therapy)
  4. Prior monoclonal antibodies, antibody-drug conjugates, or radioimmunoconjugates within 4 weeks (or 2 weeks if patient experienced disease progression on the prior treatment)
  5. Prior T-cell or other cell-based therapies within 12 weeks (or 2 weeks if patient experienced disease progression on the prior treatment)
* Part L

  1. History of radiation pneumonitis
  2. Neuropathy Grade 2 or higher
  3. Has received prior therapy with an anti-PD-1, anti-PDL1, or anti-PD-L2 agent, with an agent directed to another stimulatory or co-inhibitory T-cell receptor
  4. Has had allogenic tissue/solid organ transplant
* All Parts

  1. Recent or ongoing serious infections within 2 weeks
  2. Known positivity for hepatitis B infection
  3. Known active hepatitis C infection
  4. Active autoimmune or auto-inflammatory ocular disease within 6 months
  5. Known or suspected active organ-threatening autoimmune disease
  6. Active central nervous system tumor or metastases
* Patients with lymphomas: prior allogeneic SCT
* Patients in Part E, F, or L: history of severe immune-mediated adverse reactions or severe hypersensitivity to pembrolizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2015-02-28 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (Parts A-K) | Through 6 weeks following last dose, up to an average of 6 months
Incidence of laboratory abnormalities (Parts A-K) | Through 6 weeks following last dose, up to an average of 6 months
Objective response rate (ORR) per RECIST according to investigator assessment in the efficacy-evaluable population (Part L) | Through 6 weeks following last dose, up to an average of 6 months

SECONDARY OUTCOMES:
Incidence of adverse events (Part L) | Through 6 weeks following last dose, up to an average of 6 months
ORR per iRECIST (Part L) | Through 6 weeks following last dose, up to an average of 6 months
ORR (Parts A-K) | Through 6 weeks following last dose, up to an average of 6 months
Disease control rate (All Parts) | Through 6 weeks following last dose, up to an average of 6 months
Duration of response (All Parts) | Up to approximately 6 years
Progression-free survival (All Parts) | Up to approximately 6 years
Overall survival (All Parts) | Up to approximately 6 years
Cmax (maximum observed concentration) | Through 6 weeks following last dose, up to an average of 6 months
Tmax (time of maximum observed concentration) | Through 6 weeks following last dose, up to an average of 6 months
AUClast (AUC from time 0 to last quantifiable timepoint) | Through 6 weeks following last dose, up to an average of 6 months
AUCinf (AUC from time 0 to infinity) | Through 6 weeks following last dose, up to an average of 6 months
Apparent total clearance | Through 6 weeks following last dose, up to an average of 6 months
T1/2 (apparent terminal elimination half-life) | Through 6 weeks following last dose, up to an average of 6 months
Incidence of antitherapeutic antibodies against SEA-CD40 | Through 6 weeks following last dose, up to an average of 6 months
Blood concentrations of SEA-CD40 | Through 6 weeks following last dose, up to an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schmitt, MD, PhD, Study Director — Seagen Inc.
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - HonorHealth Scottsdale Shea Medical Center, Scottsdale, Arizona
  - Cedars Sinai Medical Center / Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Angeles Clinic and Research Institute, The, Santa Monica, California
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute / Wayne State University, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Montefiore Medical Center, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center / University of North Carolina, Chapel Hill, North Carolina
  - Case Western Reserve University / University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Seattle Cancer Care Alliance / University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Coveler AL, Smith DC, Phillips T, Curti BD, Goel S, Mehta AN, Kuzel TM, Markovic SN, Rixe O, Bajor DL, Gajewski TF, Gutierrez M, Lee HJ, Gopal AK, Caimi P, Heath EI, Thompson JA, Ansari S, Jacquemont C, Topletz-Erickson A, Zhou P, Schmitt MW, Grilley-Olson JE. Phase 1 dose-escalation study of SEA-CD40: a non-fucosylated CD40 agonist, in advanced solid tumors and lymphomas. J Immunother Cancer. 2023 Jun;11(6):e005584. doi: 10.1136/jitc-2022-005584. PMID 37385724